CLINICAL TRIAL: NCT01120457
Title: A Phase 1, Open-label, Multicenter Study of BMS-936564 (MDX-1338) in Subjects With Relapsed Acute Myelogenous Leukemia and Selected B-cell Malignancies
Brief Title: First in Human Study to Determine the Safety, Tolerability and Preliminary Efficacy of an Anti-CXCR4 Antibody in Subjects With Acute Myelogenous Leukemia and Selected B-cell Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA212-001
Record Dates: First submitted 2010-05-07; First posted 2010-05-11 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-01

CONDITIONS: Acute Myelogenous Leukemia; Diffuse Large B-Cell Leukemia; Chronic Lymphocytic Leukemia; Follicular Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular | interventions — ulocuplumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1: Dose Escalation and Expansion cohort (AML Patients) (Experimental): Dose Escalation: BMS-936564 0.3-10 mg/kg solution, Intravenous, Single 60 minute infusion as monotherapy 7 days/cycle 1 and with chemotherapy for subsequent cycles (28 days/cycle)
  Dose Expansion: BMS-936564 maximum tolerated dose (MTD) based on dose escalation, solution, Intravenous, Single 60 minute infusion as monotherapy 7 days/cycle 1 and with chemotherapy for subsequent cycles (28 days/cycle)
  Interventions: Drug: BMS-936564 (Anti-CXCR4)
- Arm 2: Dose Expansion cohort (DLBCL Patient) (Experimental): BMS-936564 MTD based on Arm 1, weekly 60 minute infusion in cycle 1 (up to 56 days) and with chemotherapy for subsequent cycles (28 days/cycle)
  Interventions: Drug: BMS-936564 (Anti-CXCR4)
- Arm 3: Dose Expansion cohort (CLL Patient) (Experimental): BMS-936564 MTD based on Arm 1, weekly 60 minute infusion in cycle 1 (up to 56 days) and with chemotherapy for subsequent cycles (28 days/cycle)
  Interventions: Drug: BMS-936564 (Anti-CXCR4)
- Arm 4: Dose Expansion cohort (FL Patient) (Experimental): BMS-936564 MTD based on Arm 1, weekly 60 minute infusion in cycle 1 (up to 56 days) and with chemotherapy for subsequent cycles (28 days/cycle)
  Interventions: Drug: BMS-936564 (Anti-CXCR4)

INTERVENTIONS:
Drug: BMS-936564 (Anti-CXCR4)
  Other Names: MDX-1338

SUMMARY:
The purpose of this study is to assess the safety and tolerability of BMS-936564 (MDX-1338) in relapsed Acute myelogenous leukemia (AML) and other selected B-cell cancers and to determine the maximum tolerated dose (MTD) of the drug alone in relapsed/refractory AML

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

A. Common to All Indications:

* Life expectancy at least 12 weeks
* ECOG Performance Status of 0-2

B. For Acute myelogenous leukemia (AML) Subjects:

* First Relapse and primary induction failure in AML (M3 excluded)
* Secondary AML subjects from myelodysplastic syndrome (MDS) or prior chemotherapy are eligible. MDS-only subjects are not eligible

C. For Follicular Lymphoma (FL), Diffuse Large B-Cell Lymphoma (DLBCL) Subjects:

* Must be at least 4 weeks (for FL) or 2 weeks (for DLBCL) since prior cytotoxic, biologic, monoclonal antibody, or investigational therapy
* Ability to undergo tumor biopsy pre-treatment and at end of monotherapy period (though not mandatory for all subjects)
* Subjects must have a histologically confirmed diagnosis of relapsed or refractory disease

D. For Chronic lymphocytic leukemia (CLL) Subjects:

* Subjects must have a histologically confirmed diagnosis of relapsed or refractory disease
* Must be at least 4 weeks since prior cytotoxic, biologic, monoclonal antibody, or investigational therapy, including corticosteroids

Exclusion Criteria:

A. Common to All indications:

* Prior anti-CXCR4 therapy including BMS-936564 (MDX-1338)
* Less than 3 months from prior hematopoietic stem cell transplant
* Presence of active graft versus host disease

B. For AML Subjects:

* Acute promyelocytic leukemia (M3)
* Left ventricular ejection fraction < institutional limits of normal

C. For FL, DLBCL Subjects:

* (For DLBCL): Inadequate renal function defined as creatinine clearance (by Cockcroft-Gault formula) < 60 mL/min
* Major surgery, not related to debulking procedures, within 21 days of first dose
* Myocardial infarction within 6 months prior to screening or Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia
* Myelodysplastic syndrome (MDS)

D. For CLL Subjects:

* No progression to more aggressive B-cell cancers, such as Richter's syndrome
* Major surgery within 21 days of Cycle 1, Day 1. Patients undergoing debulking procedures and minor surgery are allowed after a recovery period, in the judgment of the Investigator
* Myocardial infarction within 6 months prior to screening Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2010-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as monotherapy | Within the first 7 days for AML
  Safety and tolerability measured by incidence of adverse events (AEs), AEs leading to discontinuation, Serious Adverse Events (SAEs), deaths, and laboratory abnormalities
Safety and tolerability as monotherapy | Within 28 days for the selected B-cell malignancies
  Safety and tolerability measured by incidence of adverse events (AEs), AEs leading to discontinuation, Serious Adverse Events (SAEs), deaths, and laboratory abnormalities

SECONDARY OUTCOMES:
Safety, as measured by vital signs, clinical laboratory tests,ECOG performance status, physical exams, 12 lead ECGs incidence and severity of adverse events | For a maximum of thirteen 28-day cycles for the AML cohort and for a maximum of six 28-day cycles for the B-cell malignancies
  ECOG - Eastern Cooperative Oncology Group ECG - Electrocardiograms
Efficacy- including best overall response (BOR) derived from changes in tumor burden and metabolic response based on FDG-PET (for DLBCL) | For a maximum of thirteen 28-day cycles for the AML cohort and for a maximum of six 28-day cycles for the B-cell malignancies
  FDG-PET - fluoro-2-deoxyglucose positron emission tomography DLBCL - Diffuse Large B-Cell Lymphoma
Immunogenicity measurement for human anti human antibodies (HAHA) -characterizing the immunogenicity of BMS-936564 | For a maximum of thirteen 28-day cycles for the AML cohort and for a maximum of six 28-day cycles for the B-cell malignancies
  Subjects will be called as immunogenicity positive/negative to antibodies against BMS-936564 (MDX-1338) using immunogenicity assay, and will be classified as negative, positive baseline, or negative baseline with at least one positive post-treatment. The number and percentage of subjects in each classification will be reported for each dose level.
Maximum observed serum concentration (Cmax) of BMS-936564 (MDX-1338) will be derived from serum concentration versus actual time | For a maximum of thirteen 28-day cycles for the AML cohort and for a maximum of six 28-day cycles for the B-cell malignancies
Trough observed serum concentration (Cmin) of BMS-936564 (MDX-1338) will be derived from serum concentration versus actual time | For a maximum of thirteen 28-day cycles for the AML cohort and for a maximum of six 28-day cycles for the B-cell malignancies
Time of maximum observed concentration (Tmax) of BMS-936564 (MDX-1338) will be derived from serum concentration versus actual time | For a maximum of thirteen 28-day cycles for the AML cohort and for a maximum of six 28-day cycles for the B-cell malignancies
Area under the concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of BMS-936564 (MDX-1338) will be derived from serum concentration versus actual time | For a maximum of thirteen 28-day cycles for the AML cohort and for a maximum of six 28-day cycles for the B-cell malignancies
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration [AUC(0-T)] of BMS-936564 (MDX-1338) will be derived from serum concentration versus actual time | For a maximum of thirteen 28-day cycles for the AML cohort and for a maximum of six 28-day cycles for the B-cell malignancies
Area under the concentration-time curve in one dosing interval [AUC(TAU)] of BMS-936564 (MDX-1338) will be derived from serum concentration versus actual time | For a maximum of thirteen 28-day cycles for the AML cohort and for a maximum of six 28-day cycles for the B-cell malignancies
Half life (T-HALF) of BMS-936564 (MDX-1338) will be derived from serum concentration versus actual time | For a maximum of thirteen 28-day cycles for the AML cohort and for a maximum of six 28-day cycles for the B-cell malignancies
Total body clearance(CLT) of BMS-936564 (MDX-1338) will be derived from serum concentration versus actual time | For a maximum of thirteen 28-day cycles for the AML cohort and for a maximum of six 28-day cycles for the B-cell malignancies
Volume of distribution at steady-state (Vss) of BMS-936564 (MDX-1338) will be derived from serum concentration versus actual time | For a maximum of thirteen 28-day cycles for the AML cohort and for a maximum of six 28-day cycles for the B-cell malignancies
Biomarker- characterizing the pharmacodynamic (PD) profiles of BMS-936564 (MDX-1338). The main PD biomarkers are cell trafficking | For a maximum of thirteen 28-day cycles for the AML cohort and for a maximum of six 28-day cycles for the B-cell malignancies
Exploratory Biomarkers- are detection of apoptosis, cytokine analyses, CXCR4 expression, ZAP-70 and CD38 expression | For a maximum of thirteen 28-day cycles for the AML cohort and for a maximum of six 28-day cycles for the B-cell malignancies

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (11):
- United States (11):
  - Uab Comprehensive Cancer Center, Birmingham, Alabama
  - Uc San Diego Moores Cancer Center, La Jolla, California
  - Usc - Norris Comprehensive Cancer Center And Hospital, Los Angeles, California
  - Ucla-Division Of Hematology/Oncology, Los Angeles, California
  - Mayo Clinic, Jacksonville, Florida
  - Northwestern University Feinberg School Of Medicine, Chicago, Illinois
  - University Of Kansas Cancer Center And Medical Pavillion, Westwood, Kansas
  - B. Douglas Smith, M.D., Baltimore, Maryland
  - Dana-Farber Cancer Inst, Boston, Massachusetts
  - The University Of Texas Md Anderson Cancer Center, Houston, Texas
  - University Of Washington School Of Medicine, Seattle, Washington

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx